CLINICAL TRIAL: NCT06703749
Title: Simultaneous Application of HIFEM Procedure and Radiofrequency for Improvement of Muscular System Function
Brief Title: HIFEM and Radiofrequency for Muscular System Function Improvement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BTL-899_CTUS1100
Record Dates: First submitted 2024-11-19; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Muscle Damage; Muscle Strength; Muscle Weakness
Keywords: muscle; muscle impairment; lower extremities; muscle weakness
MeSH Terms: conditions — Muscle Weakness | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment with BTL-899M (Experimental): Four (4) BTL-899M treatments will be applied to the lower extremities.
  Interventions: Device: Treatment with BTL-899M
- Treatment with BTL-899M with intensities below therapeutic threshold (Placebo Comparator): Four (4) BTL-899M treatments will be applied to the lower extremities, with intensities below therapeutic threshold
  Interventions: Device: Treatment with BTL-899M with intensities below therapeutic threshold

INTERVENTIONS:
Device: Treatment with BTL-899M — The treatment administration phase will consist of four (4) treatments, delivered 5-10 days apart. The applicators of BTL-899M will be applied over the designated area. Each therapy session will last 30 minutes. The starting intensity of the radiofrequency energy will be set to 100%. The intensities of both energies will be adjusted according to the patient's feedback.
  Arms: Treatment with BTL-899M
Device: Treatment with BTL-899M with intensities below therapeutic threshold — The treatment administration phase will consist of four (4) treatments, delivered 5-10 days apart. The applicators of BTL-899M will be applied over the designated area. Each therapy session will last 30 minutes. The intensities of both energies will be set below the therapeutic threshold.
  Arms: Treatment with BTL-899M with intensities below therapeutic threshold

SUMMARY:
The goal of this clinical trial is to investigate the effect of the BTL-899M device on muscular system function in adult subjects seeking treatment for improving their muscular system function in the lower extremities. The main question it aims to answer is:

Whether the BTL-899M device is effective for muscular system function improvement 3 months posttreatment compared to the sham group, based on the dynamometer measurement.

Researchers will compare a sham group to see if the device is effective.

Participants will complete four treatment visits and two follow-up visits. Their strength will be recorded via a dynamometer.

DETAILED DESCRIPTION:
This study will evaluate the clinical efficacy and safety of the BTL-899M device for changes in muscular system function through muscle strength measurement by hand-held dynamometer. The study is a prospective, multi-center, open-label, single-arm study. The subjects will be enrolled and assigned to two groups - active and sham in a 3:1 ratio. All patients will be required to complete four (4) treatment visits receiving the treatment with the study device and two follow-up visits at 1 month and 3 months. The sham group will be treated with 5% of both energies only. The treatment administration phase will consist of four (4) treatments, delivered 5-10 days apart. The applicators of BTL-899M will be applied over the designated area. The device will induce visible muscle contractions along with heating by radiofrequency (RF). Each therapy session will last 30 minutes. At baseline, after the last treatment, and all follow-up visits, the strength measurement of the treated area will be performed by hand-held dynamometer in all subjects. At the last therapy visit, the patients will receive the Subject Satisfaction Questionnaire and Therapy Comfort Questionnaire to fill in. Subject satisfaction questionnaire will be given to the subjects at all follow-up visits. Safety measures will include documentation of adverse events (AE), which will be assessed after each procedure and at all follow-up visits. During the post-procedure visits (at 1-month and 3-month follow-up visits), all subjects will receive the Lifestyle Change Questionnaire to fill in.

ELIGIBILITY:
Inclusion Criteria:

* Age 22 years and older
* Voluntarily signed an informed consent form
* BMI ≤ 35 kg/m2
* Women of child-bearing potential are required to use birth control measures during the whole duration of the study
* Subjects willing and able to abstain from partaking in any treatments other than the pre-procedure therapy regime and the study procedure for improvement of the musculoskeletal system
* Subjects willing and able to maintain their regular (pre-procedure) diet, exercise and therapy regimen without affecting significant change in either direction during study participation

Exclusion Criteria:

* Electronic implants (such as cardiac pacemakers, defibrillators, and neurostimulators)
* Metal implants
* Drug pumps
* Malignant tumor
* Pulmonary insufficiency
* Application over muscles in the acute phase of injury
* Cardiovascular diseases
* Disturbance of temperature or pain perception
* Hemorrhagic conditions, blood coagulation disorders or anticoagulation therapy
* Septic conditions and empyema
* Acute inflammations
* Systemic or local infection such as osteomyelitis and tuberculosis
* Contagious skin disease
* Elevated body temperature
* Pregnancy, postpartum period, and nursing
* Graves' disease

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
% change from baseline in the muscle strength for the active group vs. sham group at 3 months. | baseline and 3 months
  The evaluation of the percentual (%) change in muscle strength in the active group by evaluation of dynamometer score 3 months posttreatment compared to the sham group

SECONDARY OUTCOMES:
Subject satisfaction as assessed by Subject Satisfaction Questionnaire at 3 months | from the first therapy to the 3 months after the last treatment session
  Subject Satisfaction evaluation based on the Subject Satisfaction Questionnaire administered 3 months posttreatment
Comfort as assessed by Therapy Comfort Questionnaire after the final treatment | from the first to the last treatment session, assessed up to 40 days
  Therapy comfort evaluation through the Therapy Comfort Questionnaire administered after the final treatment
Incidence of Treatment-related Adverse Events | from the first therapy to the end of subject's participation, assessed up to 5 months
  Assessment of safety throughout the course of the study by evaluting the the side effects and AE occurrence throughout the course of the study

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Royal Spine Surgery, Scottsdale, Arizona
  - The Longevity Lab, Greenwood Village, Colorado
  - Saville Spine Institute, Palm Beach Gardens, Florida